CLINICAL TRIAL: NCT02981251
Title: Effectiveness of Community Based Health Education in Reduction of Blood Pressure Among Uncontrolled Hypertensive Patients of Suburban Population of Surkhet District of Nepal
Brief Title: Community Based Health Education to Manage Uncontrolled Blood Pressure in Surkhet, Nepal
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bheri Zonal Ayurveda Hospital (Other Government)
Responsible Party: Principal Investigator, Dr. Mahesh Kumar Khanal, Director, Bheri Zonal Ayurveda Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 24/2016
Record Dates: First submitted 2016-11-30; First posted 2016-12-05 (Estimated); Last update posted 2017-09-06 (Actual); Status verified 2017-08

CONDITIONS: Hypertension
Keywords: Hypertension; Uncontrolled blood pressure; Health education; Community based
MeSH Terms: conditions — Hypertension; Health Education

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention (Experimental): Health education with support by trained female health volunteer
  Interventions: Behavioral: Health education with support by trained female health volunteer
- Control (No Intervention): Extra intervention will not be provided except usual care by their physician of the participant.

INTERVENTIONS:
Behavioral: Health education with support by trained female health volunteer — Along with usual care four sessions of interactive health education will be provided to the participants by medical officer and/or registered nurse based on a syllabus for six months. Trained female female health volunteer will motivate the participants through their home visit twice a month where they will monitor blood pressure and counsel the family members to support the patient.
  Arms: Intervention

SUMMARY:
The purpose of the study is to evaluate the effect of health education on blood pressure reduction compared to usual care among uncontrolled hypertensive patients of suburban community of Surkhet district of Nepal.

DETAILED DESCRIPTION:
Maintenance of normal blood pressure range is necessary to prevent early occurrence of cardiovascular diseases and kidney disease. Adherence of healthy behavior and lifestyle along with medication (if prescribed) are mandatory for effective management of hypertension. Although knowledge and motivation is required for such adherence through health education to the patients,however, no studies has been conducted in Nepal in community setting. Thus, our study will evaluate the effect of health education on blood pressure reduction in community settings.

Method: Cluster randomized trial will be conducted in Birendranagar Municipality of Surkhet District of Nepal. Wards will be clusters where only four ward will be selected randomly among 12 wards wards. Screening program will be conducted for uncontrolled hypertensive patients by visiting every household in systematic manner. Total 36 eligible participants will be enrolled from each cluster who meet the inclusive criteria and provide consent. Then, two clusters will be assigned to for intervention by using simple randomization procedure. Uncontrolled hypertensive patients from rest of two clusters will be the control group who will get usual care by their physician. Four sessions of hypertension related health education will be provided by medical officer and/or registered nurse to intervention group within six months. Trained female health volunteer will visit the participant's home twice a month and will record their blood pressure, motivate the patient and their family members to adhere on healthy behavior and medicine. Follow up data collection will be done after six months. Paired t- test (continues variable) and Chi-square test (binary variable) will be used to test the significance for baseline and after six months for both intervention and control group. Similarly, independent t test (continuous variable) and Chi-square test (binary variable) will be used to test the difference between the groups. Multiple logistic regression analysis will be conducted to evaluate the effect of intervention with and without adjusting confounders.

Expected Results: Primary outcome of the study will be proportion of normalized systolic blood pressure in both the groups. The study will determine the effect of intervention on the between-group difference in the proportion of patients with normalized systolic blood pressure.

Conclusion: The study will be useful to evaluate the effectiveness of health education in community setting. Thus the study will be useful for planning and implementing health education in community to control blood pressure.

ELIGIBILITY:
Inclusion Criteria:

* Who is willing to participate and give consent for the study
* Uncontrolled hypertension (SBP≥140 mmHg and/or DBP≥90mmHg) including those on antihypertensive medication
* Can understand Nepali language
* Capable of effective oral communication
* Who has telephone or mobile number -

Exclusion Criteria:

* Dementia and other mental illness
* Bed ridden patients
* Known kidney disease, cancer, heart problem, chronic obstructive pulmonary disease
* Pregnant women
* Participant who is either blind or deaf

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 142 (Actual)
Dates: Start 2016-01; Primary Completion 2017-08 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with normalized systolic blood pressure of less than 140 mm Hg | six months

SECONDARY OUTCOMES:
Proportion of patient with normal diastolic blood pressure less than 90 mm Hg | six months
Change in mean systolic and diastolic blood pressure | six months

CONTACTS AND LOCATIONS:
Overall Officials: Mahesh Kumar Khanal, MPhil, Principal Investigator — Bheri Zonal Ayurveda Hospital; Raja Ram Dhungana, MPhil, Study Director — Nepal Public Health Foundation; Yadav Gurung, MPH, Study Chair — Nepal Family Development Foundation; Pratiksha Bhandari, MA, Study Chair — Mid Western Regional Hospital; K.N. Poudel, MD, Study Chair — Surkhet Hospital Pvt. Lmt.
Locations (1):
- Bheri Zonal Ayurveda Hospital, Surkhet, Birendranagar Municipality, Nepal

IPD SHARING:
Plan to Share IPD: Undecided
Not decided yet

REFERENCES:
- [Derived] Khanal MK, Bhandari P, Dhungana RR, Bhandari P, Rawal LB, Gurung Y, Paudel KN, Singh A, Devkota S, Courten B. Effectiveness of community-based health education and home support program to reduce blood pressure among patients with uncontrolled hypertension in Nepal: A cluster-randomized trial. PLoS One. 2021 Oct 12;16(10):e0258406. doi: 10.1371/journal.pone.0258406. eCollection 2021. PMID 34637478
- [Derived] Khanal MK, Dhungana RR, Bhandari P, Gurung Y, Paudel KN. Prevalence, associated factors, awareness, treatment, and control of hypertension: Findings from a cross sectional study conducted as a part of a community based intervention trial in Surkhet, Mid-western region of Nepal. PLoS One. 2017 Oct 5;12(10):e0185806. doi: 10.1371/journal.pone.0185806. eCollection 2017. PMID 28982159